CLINICAL TRIAL: NCT02463526
Title: The Effects of Mulligan's Technique on Range of Movement, Pressure Pain Threshold, Muscle Strength, and Functionality in Subjects With Shoulder Impingement Syndrome
Brief Title: Effects of Mulligan's Technique in Subjects With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, João Flávio Guimarães, Master students, Universidade Federal de Sao Carlos
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1154-7379; 28898014.3.0000.5504 (Other: Plataforma Brasil)
Record Dates: First submitted 2015-04-30; First posted 2015-06-04 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder Impingement Syndrome; Mulligan's Mobilization with Movement; Physical Therapy
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Movement

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 - MWM condition/Sham condition (Experimental): Subjects will receive treatment for 4 times with Mulligan's Mobilization with Movement (MWM) condition, and after 72 hrs, will be treated 4 times with the sham condition.
  Interventions: Other: Mobilization with Movement (MWM) condition/ Sham condition; Other: Sham condition/ Mobilization with Movement (MWM) condition
- Group 2 - Sham condition/MWM condition (Experimental): Subjects will receive treatment for 4 times with sham condition, and after 72 hrs, will be treated 4 times with the Mulligan's Mobilization with Movement (MWM) condition.
  Interventions: Other: Mobilization with Movement (MWM) condition/ Sham condition; Other: Sham condition/ Mobilization with Movement (MWM) condition

INTERVENTIONS:
Other: Mobilization with Movement (MWM) condition/ Sham condition — The treatment condition consists in the application of a posterolateral glide (MWM) in the affected shoulder. Subjects will be seated and the therapist will stay beside the participants on the opposite side to the affected shoulder. One hand will be placed over the scapula posteriorly while the thenar eminence of the other hand will be placed over the humerus head anterior aspect. A posterior glide will be applied to the humeral head. Three sets of 10 repetitions will be applied with a 30 seconds rest interval between each set. Sham condition will replicate treatment condition except for the hand positioning. The therapist will place one hand along the clavicle and the other on the humeral head posterior aspect of the affected shoulder. A simulated anterior glide will be performed.
Other: Sham condition/ Mobilization with Movement (MWM) condition — The Sham condition consists in the application of a simulated anterior glide in the affected shoulder. Subjects will be seated and the therapist will stay beside the participants on the opposite side to the affected shoulder. The therapist will place one hand along the clavicle and the other on the humeral head posterior aspect of the affected shoulder. A simulated anterior glide will be performed. Three sets of 10 repetitions will be applied with a 30 seconds rest interval between each set. The treatment condition will replicate treatment condition except for the hand positioning. The therapist will place one hand over the scapula posteriorly while the thenar eminence of the other hand will be placed over the anterior humerus head. A posterior glide will be applied to the humeral head.

SUMMARY:
Participants will be initially assessed for their suitability for inclusion in the study and will undergo a physical screening of the affected shoulder and cervical spine by an experienced physiotherapist. After, participants will be attended 72 hours after data recording of the baseline measures (range of motion with a goniometer, pressure pain threshold with a algometer, and peak force with a dynamometer) for four sessions per week with 24 hours of interval between sessions. At each experimental week session, each participant will receive one of the two treatment conditions (MWM or sham) and then will repeats the assessment. In the following week, there will be a crossover condition of each individual and 24 hours after the last treatment session, the examiner will do the last assessment.

ELIGIBILITY:
Inclusion Criteria:

* history of shoulder pain of >1-week duration, localized at the proximal anterolateral shoulder region consistent to Shoulder Impingement Syndrome (SIS);
* at least 1 positive impingement test (Jobe's test, Neer's test, Hawkins-Kennedy's Test) associated with painful range of motion during arm elevation; or pain during external rotation with the arm in 90 degrees of elevation in the coronal plane.

Exclusion Criteria:

* fibromyalgia (based on self-report),pregnancy, a history of onset of symptoms because of traumatic injury, other histories of shoulder injury, torn tendons, ligamentous laxity based on positive Sulcus test and apprehension test, numbness or tingling in the upper extremity, previous shoulder or neck surgery, systemic illnesses, body mass index > 28kg/m2, corticosteroid injection 3 months before evaluation, physical therapy 3 months before evaluation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pressure Pain Threshold | 72 hours before the treatment starts, 24 hours after the last MWM or Shaw treatment, and 24 hours after the last treatment.
  The pressure pain threshold will be assessed with a algometer and the unit of measure is the kilogram per square centimeter.

SECONDARY OUTCOMES:
Range of Motion | 72 hours before the treatment starts, 24 hours after the last MWM or Shaw treatment, and 24 hours after the last treatment.
  The range of motion will be assessed with a goniometer and the unit of measure is the degree
Peak Force | 72 hours before the treatment starts, 24 hours after the last MWM or Shaw treatment, and 24 hours after the last treatment.
  The Peak Force will be assessed with a handheld dynamometer and the unit of measure is the kilogram.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Alburquerque-Sendín, Professor, Study Director — Universidade Federal de Sao Carlos; Tania Salvini, Professor, Study Chair — Universidade Federal de Sao Carlos
Locations (1):
- UFSCar, São Carlos, São Paulo, Brazil